CLINICAL TRIAL: NCT00266656
Title: Effect of Early Growth Hormone Treatment on Long-term Growth and Skeletal Maturation in Girls With Turner Syndrome
Brief Title: Long-Term Growth and Skeletal Effects of Early Growth Hormone Treatment in Turner Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10088; B9R-US-GDGH (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental 1 Control (Experimental): No drug administration in B9R-US-GDFG (NCT00406926).
  Humatrope according to investigator's clinical practice and guided by the approved package insert on whether treatment is given.
  Interventions: Drug: Humatrope
- Experimental 2 Humatrope (Experimental): Humatrope according to investigator's clinical practice and guided by the approved package insert on whether treatment is given.
  Interventions: Drug: Humatrope

INTERVENTIONS:
Drug: Humatrope — According to investigator's clinical practice and guided by the approved package insert
  Other Names: LY137998; Somatropin; Growth hormone

SUMMARY:
This is an extension study that will gather long-term data on the effect of early growth hormone (GH) treatment on adult height and other aspects of health and development in girls with Turner syndrome. The main purpose is to determine whether girls who received 2 years of GH treatment before 6 years of age achieve taller adult height than girls who were untreated during this time. The study will also look at middle ear and hearing function, and cognitive and behavioral development. Protocol completion is defined as attainment of height velocity less than or equal to 1.0 cm/year, or bone age greater than or equal to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously randomized in study B9R-US-GDFG (NCT00406926)
* Karyotype-proven Turner syndrome

Exclusion Criteria:

* Immediate family members of study site personnel directly affiliated with the study

Ages: 4 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2005-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hrs), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Hospital of Chicago Research Center, Chicago, Illinois
  - Riley Hosptial for Children, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of NC at Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Childrens Hospital and Medical Center, Seattle, Washington

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To be included in this study, participants had to be females with karyotype-proven Turner syndrome who were previously randomized in Study B9R-US-GDFG (NCT00406926).
Groups:
- Early Treated: Humatrope administered according to investigator's clinical practice and guided by the approved package insert.
  Humatrope administered in B9R-US-GDFG (NCT00406926).
- Early Untreated: Humatrope administered according to investigator's clinical practice and guided by the approved package insert.
  Control: Humatrope was not administered in B9R-US-GDFG (NCT00406926).
Period: Overall Study
Arm/Group | Early Treated | Early Untreated
Started | 36 | 33
Completed | 22 | 20
Not Completed | 14 | 13
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Did Not Reach Final Height | 4 | 8
Not completed — Parent/Caregiver Decision | 1 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled/started participants.
Groups:
- Early Treated: Early treated n=36
- Early Untreated: Early untreated n=33
- Total: Total of all reporting groups
Arm/Group | Early Treated | Early Untreated | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.29 (1.22) | 8.41 (1.30) | 8.35 (1.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeter] | 124.34 (10.08) | 121.06 (9.76) | 122.77 (9.99)
Height Standard Deviation Score (SDS) [Mean (Standard Deviation); unit: Standard Deviation Score] | -0.84 (1.22) | -1.48 (1.23) | -1.15 (1.26)
Bone Age [Mean (Standard Deviation); unit: years] | 8.73 (1.55) | 8.34 (1.57) | 8.54 (1.56)

OUTCOME MEASURES:

1. Primary Outcome: Most Mature Height Standard Deviation Score (SDS)
Description: SDS reports the number of standard deviations from the mean for age and sex for an individual measurement (normal range is -2 to +2 SDS). Height SDS is derived by subtracting the population mean from individual's height value and then dividing that difference by the population standard deviation. Greater height SDS values indicate greater height.
Time Frame: Baseline through End of Study (10 years)
Population: All participants who achieved Near Adult Height (NAH). NAH is defined as first height measured when height velocity is less than or equal to 2.0 centimeter per year over the preceding year (in the absence of growth-impairing process such as hypothyroidism or inflammatory bowel disease), or bone age greater than or equal to14.5 years.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 25 | 26
standard deviation score | -1.37 (1.09) | -1.60 (1.21)

2. Secondary Outcome: Height SDS at Various Ages
Description: as for outcome 1
Time Frame: Age 10, Age 13, Age 16
Population: All participants who had a baseline visit and at least one post-baseline visit.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 35 | 32
Standard deviation score
  Age 10 (n=32, 30) | -0.66 (1.16) | -1.28 (1.17)
  Age 13 (n=29, 29) | -1.29 (1.24) | -1.87 (1.16)
  Age 16 (n=18, 18) | -1.66 (1.11) | -1.69 (1.30)

3. Secondary Outcome: Age at Attainment of Tanner 2 Breast Development
Description: The Tanner 2 breast development is the age at first evidence of breast development.
Time Frame: Baseline through End of Study (10 years)
Population: All participants who had a baseline visit and at least one post-baseline visit.
Measure: Mean (Standard Error); unit: years
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 35 | 32
years | 11.80 (0.26) | 12.14 (0.31)

4. Secondary Outcome: Chronological Age at First Visit Participant Attained Bone Age of 14.5 Years
Description: Bone age was measured by standard radiograph, x-ray at baseline and annually for 10 years or until attainment of height velocity less than or equal to 1.0 centimeter per year (cm/year) and bone age greater or equal to 15 years.
Time Frame: Baseline through End of Study (10 years)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: years
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 25 | 26
years | 14.64 (0.25) | 15.26 (0.23)

5. Secondary Outcome: Reports of Serious Adverse Events
Description: Number of serious adverse events (SAEs) reported. Any adverse event from this study that results in one of the following outcomes, or is significant for any other reason were reported as an SAE: death, initial or prolonged inpatient hospitalization, a life-threatening experience (that is, immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect in the offspring of a study subject, significant for any other reason (includes cancer, other than superficial, and basal cell or squamous cell carcinomas of the skin, that did not meet other serious adverse event criteria).
  A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through End of Study (10 years)
Population: All participants who had a baseline visit, regardless of whether or not they received Humatrope at any time.
Measure: Number; unit: events
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 36 | 33
events | 8 | 5

6. Secondary Outcome: Percentage of Participants With Occurrence of Pre-specified Clinically Relevant Events
Description: Percentage of participants for whom certain non-serious, pre-specified adverse events (AEs; those that are commonly observed in Turner syndrome or are known to be related to GH treatment: impaired glucose tolerance, diabetes mellitus, hypothyroidism, benign intracranial hypertension, scoliosis, slipped capital femoral epiphysis, solid tumor/leukemia, pancreatitis, ear infections, and high blood pressure) are reported.
Time Frame: Baseline through End of Study (10 years)
Population: All participants who had a baseline visit, regardless of whether or not they received Humatrope at any time.
Measure: Number; unit: percentage of participants
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 36 | 33
percentage of participants
  Baseline Ear infections | 13.9 | 18.2
  Baseline High Blood Pressure | 0 | 3.0
  Baseline Hypothyroidism | 13.9 | 6.1
  Baseline Scoliosis | 22.2 | 9.1
  Year 1 Ear infections | 38.9 | 39.4
  Year 1 High Blood Pressure | 0 | 3.0
  Year 1 Hypothyroidism | 11.1 | 12.1
  Year 1 Scoliosis | 16.7 | 21.2
  Year 2 Diabetes | 2.8 | 0
  Year 2 Dilatation of the Aorta | 0 | 3.0
  Year 2 Ear infections | 33.3 | 27.3
  Year 2 High Blood Pressure | 0 | 3.0
  Year 2 Hypothyroidism | 11.1 | 12.1
  Year 2 Scoliosis | 22.2 | 24.2
  Year 3 Diabetes | 2.8 | 0
  Year 3 Dilatation of the Aorta | 0 | 6.1
  Year 3 Ear infections | 30.6 | 36.4
  Year 3 High Blood Pressure | 0 | 3.0
  Year 3 Hypothyroidism | 11.1 | 12.1
  Year 3 Scoliosis | 25.0 | 27.3
  Year 4 Diabetes | 2.8 | 0
  Year 4 Dilatation of the Aorta | 0 | 6.1
  Year 4 Ear infections | 16.7 | 30.3
  Year 4 High Blood Pressure | 0 | 3.0
  Year 4 Hypothyroidism | 11.1 | 12.1
  Year 4 Scoliosis | 25.0 | 27.3
  Year 5 Diabetes | 2.8 | 0
  Year 5 Dilatation of the Aorta | 0 | 6.1
  Year 5 Ear infections | 22.2 | 27.3
  Year 5 High Blood Pressure | 0 | 3.0
  Year 5 Hypothyroidism | 13.9 | 18.2
  Year 5 Scoliosis | 25.0 | 27.3
  Year 6 Diabetes | 2.8 | 0
  Year 6 Dilatation of the Aorta | 0 | 9.1
  Year 6 Ear infections | 19.4 | 24.2
  Year 6 High Blood Pressure | 0 | 3.0
  Year 6 Hypothyroidism | 13.9 | 18.2
  Year 6 Scoliosis | 16.7 | 30.3
  Year 7 Diabetes | 2.8 | 0
  Year 7 Dilatation of the Aorta | 0 | 9.1
  Year 7 Ear infections | 19.4 | 18.2
  Year 7 High Blood Pressure | 0 | 3.0
  Year 7 Hypothyroidism | 13.9 | 15.2
  Year 7 Scoliosis | 13.9 | 30.3
  Year 8 Diabetes | 2.8 | 0
  Year 8 Dilatation of the Aorta | 2.8 | 9.1
  Year 8 Ear infections | 13.9 | 18.2
  Year 8 High Blood Pressure | 0 | 3.0
  Year 8 Hypothyroidism | 5.6 | 12.1
  Year 8 Scoliosis | 13.9 | 33.3
  Year 9 Dilatation of the Aorta | 0 | 3.0
  Year 9 Ear infections | 2.8 | 3.0
  Year 9 High Blood Pressure | 0 | 3.0
  Year 9 Hypothyroidism | 2.8 | 6.1
  Year 9 Scoliosis | 5.6 | 9.1
  Year 10 Scoliosis | 2.8 | 0

7. Secondary Outcome: Percentage of Participants With Abnormal Tympanometry Results
Description: Percentage of participants with abnormal tympanometry [defined as middle ear dysfunction / middle ear effusion / patent pressure equalizer tube or possible tympanic membrane perforation] results at baseline, age 10 years, and age 16 years or endpoint.
Time Frame: Baseline, Age 10, Age 16, End of Study (10 years)
Population: All participants who had a baseline visit, regardless of whether or not they received Humatrope at any time.
Measure: Number; unit: percentage of participants
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 36 | 33
percentage of participants
  Baseline Right Ear | 44.4 | 54.5
  Baseline Left Ear | 47.2 | 45.5
  Age 10 Right Ear | 27.8 | 15.2
  Age 10 Left Ear | 27.8 | 15.2
  Age 16 Right Ear | 2.8 | 9.1
  Age 16 Left Ear | 2.8 | 3.0
  Endpoint Right Ear | 8.3 | 12.1
  Endpoint Left Ear | 11.1 | 9.1

8. Secondary Outcome: Percentage of Participants With Prevalence of Abnormal Audiometry Results
Description: Percentage of participants with abnormal Audiometry results at baseline, age 10 years, and age 16 years or endpoint. Prevalence was calculated as number of participants with abnormal hearing divided by number of participants with measurable pure tone audiometry results at that visit.
Time Frame: Baseline, Age 10, Age 16, End of Study (10 years)
Population: All participants who had a baseline visit, regardless of whether or not they received Humatrope at any time.
Measure: Number; unit: percentage of participants
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 36 | 33
percentage of participants
  Baseline Visit (n=36, 33) | 52.8 | 48.5
  Age 10 (n=27, 24) | 44.4 | 29.2
  Age 16 (n=7, 9) | 85.7 | 66.7
  Endpoint (n=24, 22) | 37.5 | 40.9

9. Secondary Outcome: Percentage of Participants With Abnormal Audiometry Results Based on Pure Tone Average (PTA)
Description: Percentage of participants with abnormal Audiometry results at baseline, age 10 years, and age 16 years or endpoint. PTA is defined as the average of pure tone hearing thresholds at 500, 1000 and 2000 Hz (Hertz), calculated separately for each ear and for each testing method (air or bone); normal PTA is defined as pure tone hearing threshold less than or equal to 20 dB HL (decibels Hearing Level), and abnormal PTA is defined as pure tone hearing threshold greater than 20 DB HL.
Time Frame: Baseline, Age 10, Age 16, End of Study (10 years)
Population: All participants who had a baseline visit, regardless of whether or not they received Humatrope at any time.
Measure: Number; unit: percentage of participants
Arm/Group | Early Treated | Early Untreated
Number analyzed (Participants) | 36 | 33
percentage of participants
  Baseline Left Ear Air (n=36, 32) | 30.6 | 31.3
  Baseline Left Ear Bone (n=36, 32) | 2.8 | 0.0
  Baseline Right Ear Air (n=36, 32) | 22.2 | 37.5
  Baseline Right Ear Bone (n=36, 32) | 22.2 | 2.8
  Age 10 Left Ear Air (n=27, 21) | 29.6 | 14.3
  Age 10 Left Ear Bone (n=27, 21) | 0.0 | 0.0
  Age 10 Right Ear Air (n=27, 22) | 14.8 | 18.2
  Age 10 Right Ear Bone (n=27, 22) | 0.0 | 9.1
  Age 16 Left Ear Air (n=7, 9) | 57.1 | 66.7
  Age 16 Left Ear Bone (n=7, 9) | 0.0 | 0.0
  Age 16 Right Ear Air (n=7, 9) | 28.6 | 33.3
  Age 16 Right Ear Bone (n=7, 9) | 0.0 | 22.2
  Endpoint Left Ear Air (n=20, 20) | 30.0 | 35.0
  Endpoint Left Ear Bone (n=20, 20) | 5.0 | 20.0
  Endpoint Right Ear Air (n=20, 20) | 20.0 | 35.0
  Endpoint Right Ear Bone (n=20, 20) | 10.0 | 25.0

ADVERSE EVENTS:
Description: All enrolled/started participants.
Arm/Group | Early Treated | Early Untreated
Serious Adverse Events (participants affected / at risk) | 6/36 | 5/33
Other Adverse Events (participants affected / at risk) | 34/36 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Treated (N=36) | Early Untreated (N=33)
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pterygium colli (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early Treated (N=36) | Early Untreated (N=33)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 4 (4) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 6 (8) | 3 (4)
Hearing impaired (Ear and labyrinth disorders) | 2 (2) | 3 (3)
Tympanic membrane perforation (Ear and labyrinth disorders) | 7 (8) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 5 (5)
Myopia (Eye disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Tooth malformation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (12) | 3 (3)
Pain (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 11 (11) | 8 (8)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Multiple allergies (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 5 (5) | 2 (2)
Bronchitis (Infections and infestations) | 5 (5) | 4 (4)
Conjunctivitis (Infections and infestations) | 4 (4) | 3 (3)
Croup infectious (Infections and infestations) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 7 (7) | 2 (2)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 4 (5)
Impetigo (Infections and infestations) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 3 (3)
Kidney infection (Infections and infestations) | 2 (2) | 0 (0)
Mononucleosis syndrome (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (9) | 4 (5)
Otitis externa (Infections and infestations) | 3 (4) | 5 (6)
Otitis media (Infections and infestations) | 9 (11) | 12 (14)
Pharyngitis streptococcal (Infections and infestations) | 4 (4) | 9 (9)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 7 (7) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (7)
Urinary tract infection (Infections and infestations) | 8 (9) | 0 (0)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 4 (5) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Echocardiogram normal (Investigations) | 2 (2) | 6 (6)
Electrocardiogram normal (Investigations) | 1 (1) | 2 (2)
Ultrasound kidney normal (Investigations) | 2 (2) | 2 (2)
Ultrasound scan normal (Investigations) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (10)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 9 (9)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 4 (4)
Headache (Nervous system disorders) | 11 (13) | 9 (10)
Anxiety (Psychiatric disorders) | 7 (7) | 6 (6)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Enuresis (Renal and urinary disorders) | 1 (1) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Corrective lens user (Social circumstances) | 3 (3) | 8 (8)
Orthodontic appliance user (Social circumstances) | 9 (9) | 7 (7)
Adenoidectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Ear tube insertion (Surgical and medical procedures) | 4 (5) | 5 (7)
Mole excision (Surgical and medical procedures) | 6 (6) | 2 (2)
Oral surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Orthodontic procedure (Surgical and medical procedures) | 4 (4) | 7 (7)
Palatal operation (Surgical and medical procedures) | 3 (3) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 2 (2)
Tympanoplasty (Surgical and medical procedures) | 5 (5) | 3 (3)
Wisdom teeth removal (Surgical and medical procedures) | 2 (2) | 1 (1)
Aortic dilatation (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Lymphoedema (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days